CLINICAL TRIAL: NCT05770219
Title: Expanded Access Program: TAK-755 (rADAMTS13) for the Prophylaxis and Treatment of Severe Congenital or Hereditary Thrombotic Thrombocytopenic Purpura
Brief Title: Expanded Access Program of TAK-755 for Congenital Thrombotic Thrombocytopenic Purpura (cTTP)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-755 EAP
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
Keywords: Drug Therapy
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: TAK-755 — TAK-755 as IV injection at dose calculated based on the participant's body weight as measured at each dosing visit. For most participants, the final volume of infusion will be between 5 and 14 mL.
  Other Names: recombinant ADAMTS13 (rADAMTS13)

SUMMARY:
The expanded access program allows people to gain access to unlicensed treatment on compassionate grounds. TAK-755 also known as rADAMTS13, is a medicine that treats people born with severe congenital or hereditary thrombotic thrombocytopenic purpura (cTTP). This expanded access program enables continued access to those participants who have no other treatment options available for cTTP.

DETAILED DESCRIPTION:
This is an expanded access program in which the drug being given is called TAK-755. This study will provide access to TAK-755 prior to marketing authorization for eligible participants with severe congenital or hereditary TTP who cannot adequately be treated via current standard of care and who cannot enter a clinical trial.

All participants will receive TAK-755 as intravenous (IV) injection based on their weight as measured at each dosing visit.

This is a multi-center, international program. Participants will continue treatment until benefit is no longer derived from the treatment (or treatment is no longer tolerable), sponsor decision, the participant chooses to discontinue the treatment, or TAK-755 becomes commercially available.

ELIGIBILITY:
Inclusion Criteria:

1. Participant or legally authorized representative has provided signed informed consent (≥18 years of age) and/or assent form (signed by legal representative if participants is <18 years of age).
2. Participant has a documented diagnosis of severe congenital ADAMTS13 deficiency, defined by:

   1. Confirmed molecular genetic testing, or
   2. ADAMTS13 activity and a negative test for ADAMTS13 antibodies.
3. Participant is currently on a prophylactic regimen or has a documented history of at least 1 TTP event.
4. Standard of Care (SoC) is considered inadequate, or the participant is intolerant to SoC*.

   * SoC are plasma-based therapies, e.g., fresh frozen plasma or S/D treated plasma

Exclusion Criteria:

1. Participant is currently eligible to enter into an interventional clinical trial for cTTP.
2. There is a suitable alternative commercially available treatment for the treatment of cTTP.
3. Participant has been diagnosed with any other thrombotic microangiopathies (TMAs) like disorder (microangiopathic hemolytic anemia), including acquired TTP.
4. Participant has a known hypersensitivity/allergies/intolerance or contraindications to TAK-755 or its excipients, such as hamster proteins.
5. Participant has a medical history or presence of a functional ADAMTS13 inhibitor.
6. Participant has a medical history of genetic or acquired immune deficiency that would interfere with the assessment of product immunogenicity, including Participants who are human immunodeficiency virus (HIV)-positive with an absolute cluster of differentiation 4 (CD4) count <200 per millimeter cube (<200/mm^3) or who are receiving chronic immunosuppressive drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- See also: To obtain more information on the study, click here on this link — https://clinicaltrials.takeda.com/study-detail/4e6348797ec74b0a?idFilter=%5B%22TAK-755+EAP%22%5D